CLINICAL TRIAL: NCT03832127
Title: Exploratory Study Evaluating the Interest of PET to 18F-Fludarabine for the Initial Assessment and End-treatment Evaluation of Patients With Symptomatic Multiple Myeloma in the First Line of Treatment, Not Candidates for Marrow Autograft
Brief Title: Evaluation of PET 18F-Fludarabine for the Initial Assessment and End-treatment of Symptomatic Multiple Myeloma Patients
Acronym: Myelofludate
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Cyceron (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC18_0055
Record Dates: First submitted 2018-07-20; First posted 2019-02-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludatep (Experimental): PET with 18F-Fludarabine
  Interventions: Drug: 18F-Fludarabine

INTERVENTIONS:
Drug: 18F-Fludarabine — Two PET with 18F-Fludarabine : one at Baseline, the second one at the end of treatment of myeloma

SUMMARY:
The objective of this exploratory study is to evaluate, for the first time, the sensitivity of 18F-Fludarabine to the initial diagnosis of MM compared to FDG-PET and MRI. The interest of this molecule will also be investigated as part of the end-of-treatment therapeutic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic MM in the first line in patients who are not candidates for autologous bone marrow transplantation.
* Patients eligible for one of the treatments considered as standard in a patient who is not eligible for autograft, according to ESMO's European recommendations
* MM with measurable disease either by the serum evaluation of the monoclonal component or by the determination of free light chains (serum or urinary).
* Patient affiliated with a social insurance scheme
* The patient must understand and voluntarily sign the informed consent form
* Women of childbearing potential must have a serum pregnancy test (performed within 2 days before each PET scan.)
* Women of childbearing potential must use an effective contraceptive method throughout the course of the study and for 30 days after the last PET.
* Male patients (vasectomised or not) with a pregnant partner or a partner of childbearing potential must use a condom and a spermicide until 90 days after the last PET.
* HIV serology known to be negative
* Karnofsky ≥ 70 or ECOG 0-1

Exclusion Criteria:

* Age under 18 years
* Pregnancy or breastfeeding
* Male or female refusing birth control conditions
* Primary AL amyloidosis and myeloma complicated by amyloidosis
* Neutropenia <1000 PN / mm3
* Thrombocytopenia <70,000 / mm3
* Hepatic impairment: bilirubin> 35μmol / L and SGOT, SGPT, alkaline phosphatase greater than 3 N
* Renal impairment defined by creatinine clearance <50 ml / min
* History of other malignancies with the exception of basal cell carcinoma and stage I cervical cancer
* Severe active infection
* Active infection with known hepatitis B or C virus.
* Patient with insulin-dependent or non-insulin-dependent diabetes mellitus.
* Intolerance or known allergy to any of the study drugs or any of its analogues
* Psychiatric illness that may interfere with participation in the study
* Patient under safeguard of justice
* Intellectual inability to sign informed consent
* Persons protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-09-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Detection of sensitivity of the lesions (osseous and extra-osseous) of 18Fludarabine PET (FludaTEP) | Before treatment
  The sensitivity of the initial FludaTEP will be evaluated using an optimal reading mode lesion analysis (ie by consensus of experts) by defining :
  True positive:
  * positive lesion with 18F-Fludarabine and positive with PET-FDG or MRI
  * or positive lesion with 18-F-Fludarabine, negative with PET-FDG and MRI, but confirmed by further complementary imaging (CT) or histological examination, or confirmed at follow-up
  False negative:
  -negative lesion with 18F-Fludarabine and positive FDG-PET and / or MR Lesions positivity in PET-FDG and MRI will be assessed by central reading done by consensus of experts. Lesions positivity with 18F-Fludarabine will be defined by central reading assessed by 2 nuclear physicians experts in hematology with no access to the other exams' results.

SECONDARY OUTCOMES:
To evaluate the specificity and the positive and negative predictive values of the FludaTEP for the initial assessment through an optimal reading mode. | Before treatment
  The specificity, positive predictive value (PPV) and negative predictive value (NPV) of the FludaTEP for the initial assessment will be assessed through an optimal reading mode lesion analysis (ie by consensus of experts) using same true positive and false positive définitions as for the main endpoint and defining: -positive lesion with 18F-Fludarabine but not found or confirmed on an histological examination, or other imaging technique (PET-FDG, MRI +/- Scan) or at follow-up
  True negative:
  -negative lesion with 18F-Fludarabine and negative with FDG-PET and MRI
To evaluate the sensitivity, specificity, and positive and negative predictive values of the FludaTEP for the initial balance according to the local reading | Before treatment
  The specificity, positive predictive value (PPV) and negative predictive value (NPV) of the FludaTEP for the initial balance will be evaluated through lesion analysis based on the local reading investigator center reading using definitions of VP, VN, FP, and FN described above.
To evaluate the prognostic impact of FDG-PET and FludaTEP on the number of lesions detected by each imaging technique in a population of MM patients in the 1st line therapeutic but not candidates for marrow autograft. | After treatment
  The prognostic impact of FDG-PET and FludaTEP as a function of the number of lesions detected by each imaging technique will be evaluated by evaluating the impact of these data on progression-free survival and overall survival. Progression-free survival is defined as the time between the beginning of treatment of the disease and relapse or progression. Overall survival is defined as the time between the start of treatment and death.
To evaluate the prognostic impact of FludaTEP on the initial assessment and for the end-of-treatment therapeutic evaluation | Before and After treatment
  The prognostic impact of FludaTEP on the initial assessment and for the end-of-treatment therapeutic evaluation will be determined by evaluating the impact of a decrease and a negation of the signal in imaging on an increase in progression-free survival and overall survival.
Evaluate in a population of MM patients the existence of a correlation between the 18Fludarabine and FDG uptake intensities | Before and After treatment
  Correlations between the 18Fludarabine and FDG uptake intensities assessed by SUVs and the quantitative expression of markers measured in flow cytometry and cytogenetic data (in particular the expression of the coding gene for hexokinases) will be measured using Spearman's correlation coefficient.
Evaluate in a population of MM patients the existence of a correlation between the 18Fludarabine and FDG uptake intensities and the cytogenetic data Tolerance to 18F-Fludarabine | Before and After treatment
  Tolerance to 18F-Fludarabine will be evaluated by clinical monitoring during 2 hours following the 18F-Fludarabine injection. Clinical data will be taken prior to the 18F-Fludarabine injection, prior to the data capture at 60min and after the last data capture.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CHU de Nantes, Nantes
  - Centre Eugène Marquis, Rennes
  - CHU de Rennes, Rennes
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided